CLINICAL TRIAL: NCT05288725
Title: A Study to Evaluate the Safety, and Efficacy of Minimally Manipulated Autologous Bone Marrow Aspirate to Treat Knee Osteoarthritis in Patients
Brief Title: Mesenchymal Stem Cell Therapy for Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Next Generation Regenerative Medicine LLC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGRM-001
Record Dates: First submitted 2022-02-15; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Osteoarthritis; Knee Pain; Bone Marrow Aspirate; Mesenchymal Stem Cells; Cell Therapy; Corticosteroid; Regenerative Medicine; Functional Improvement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Adrenal Cortex Hormones; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Corticosteroid as control both participant and investigator blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Intra-articular injection with Bone Marrow Derived Mesenchymal Stem Cells (MSCs) (Experimental): Participants will undergo a bone marrow aspirate procedure. Participants will receive a single intra-articular injection of NGRM-001 on treatment day.
  Interventions: Biological: Bone Marrow Derived MSCs; Device: Bone Marrow Aspirate
- Subchondral injection with Bone Marrow Derived MSCs (Experimental): Participants will undergo a bone marrow aspirate procedure. Participants will receive a single subchondral injection of NGRM-001 on treatment day.
  Interventions: Biological: Bone Marrow Derived MSCs; Device: Bone Marrow Aspirate
- Combined Intra-articular and Subchondral injection with Bone Marrow Derived MSCs (Experimental): Participants will undergo a bone marrow aspirate procedure. Participants will receive a single combined intra-articular and subchondral injection of NGRM-001 on treatment day.
  Interventions: Biological: Bone Marrow Derived MSCs; Device: Bone Marrow Aspirate
- Corticosteroid injection (Active Comparator): Subjects in the corticosteroid group will undergo a mock bone marrow aspirate procedure. Participants will receive a single intra-articular injection of corticosteroid on treatment day.
  Interventions: Drug: Corticosteroid; Device: Bone Marrow Aspirate

INTERVENTIONS:
Biological: Bone Marrow Derived MSCs — Autologous bone marrow aspirate (BMA) is an orthobiologic injection used in knee osteoarthritis therapy. Bone marrow aspirate is harvested from the posterior superior iliac crest (PSIS) of the spine using the Marrow Cellutions kit. BMA will be injected into the knee using ultrasound guidance.
  Other Names: Bone Marrow Aspirate; Marrow Cellutions
  Arms: Combined Intra-articular and Subchondral injection with Bone Marrow Derived MSCs; Intra-articular injection with Bone Marrow Derived Mesenchymal Stem Cells (MSCs); Subchondral injection with Bone Marrow Derived MSCs
Drug: Corticosteroid — The corticosteroid is prepared in a 10 ml syringe by combining 1-2 mL Kenalog [40 mg/dL], 6-8 mL sterile normal saline, 3-4 mL Ropivicaine 1%.
  Other Names: Kenalog
  Arms: Corticosteroid injection
Device: Bone Marrow Aspirate — The Marrow Cellutions kit is an FDA approved device for harvesting bone marrow aspirate.

SUMMARY:
The study is a multicentered, randomized, double-blinded, placebo-controlled study conducted on the unilateral knee of 120 patients. The study compares the effectiveness of an injection of a mesenchymal stem cell preparation from autologous bone marrow aspirate (BMA) to a corticosteroid control for knee osteoarthritis. WOMAC, VAS pain scores, and MRI will be used for assessment. The study will be conducted at 3 sites in the United States.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis in the knee that affects millions of adults throughout the world and is the leading cause of disability. It is a degenerative type of arthritis that occurs most often in patients, as the cartilage in the knee joint gradually wears away. As the cartilage wears away, it becomes frayed and rough, and the protective space between the bones decreases. This can result in bone rubbing on bone and produce painful bone spurs. The patient experiences pain that worsens over time.

Although current surgical therapeutic procedures to cartilage repair are clinically useful, they cannot restore a normal articular surface, and in many cases, resulted in the growth of inferior quality fibrocartilage. Therefore, techniques and practices have been developed to collect minimally manipulated bone marrow aspirate (BMA), that contains Bone Marrow Derived Mesenchymal Stem Cells (BMDMSCs) and other endogenous acellular components, from knee OA patients for autologous transplantation in the treatment of their knee OA.

Participants will be randomized to study arms to receive a BMA injection to the intra-articular knee, subchondral knee, both intra-articular and subchondral knee, or to receive a corticosteroid injection to the knee. A corticosteroid injection is currently the standard of care for osteoarthritis patients having knee pain. All participants will undergo a procedure. Participants will be blinded as to whether they receive a BMA injection or a corticosteroid injection.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be willing and able to provide written informed consent.
2. Healthy, non-smoking, males and females.
3. Negative Pregnancy test.
4. Body weight > 45 kg and Body Mass Index (BMI) between 18 and 40 kg/m2 (i.e., subjects with a BMI >40 and <18 will be excluded).
5. No clinically significant abnormal findings on blood pressure, heart rate, physical examination, clinical laboratory tests, or Electrocardiogram (ECG). See details below:

   1. Heart Rate (HR) >60 and <100 bpm
   2. Systolic Blood Pressure (BP) >90 and <170 mmHg
   3. Diastolic BP >60 and <80 mmHg
   4. Pulse oximetry ≥95% at room air
   5. Temperature: normal
   6. Laboratory measures within normal range
   7. Liver enzymes <2 x Upper Limit of Normal (ULN)
   8. Normal bilirubin
   9. Normal Pain Threshold (PT) / International Normalized Ratio (INR)
   10. Estimated Glomerular Filtration Rate (eGFR) >60 ml/min
   11. Normal ECG.
6. Individuals 18 to 80 years old that have knee Osteoarthritis.
7. X-rays that demonstrate OA with the Kellgren-Lawrence grading scale of 2, 3 or 4 in at least one compartment of the knee either or both knees. Only subjects that have a single symptomatic knee will be enrolled.
8. No significant Medial Collateral Ligament (MCL) or Lateral Collateral Ligament (LCL) tear or laxity. (A significant LCL and MCL laxity or tear would be determined on clinical exam if there is no endpoint on valgus or Varus stress physical exam. Upon review of the MRI, NGRM will only treat subjects with no grade 2 or grade 3 ligamentous sprains [LCL, MCL, Anterior Cruciate Ligament (ACL), Posterior Cruciate Ligament (PCL)]. Next Generation Regenerative Medicine (NGRM) will treat subjects with degenerative meniscal changes in tears but no acute or large bucket handle tears.)
9. No significant meniscal tear. (i.e. bucket handle) (A positive McMurrays test on clinical exam indicates a significant meniscal tear. The subjects will also be getting a baseline MRI that will help delineate any further ligament injuries that may disqualify a subject.)
10. Subjects who have had the benefit of standard of care (SOC) treatment (activity modification, weight loss, physical therapy, anti-inflammatory medications, or injection therapy) before receiving experimental therapy. However, subjects cannot have had the benefit of standard of care treatment at less than 3 months before receiving experimental therapy. Enroll subjects who have demonstrated failure or are intolerant to SOC treatment. The time frame prior to screening when failure of conservative treatment would have occurred will be one year of symptoms and failure of conservative treatment which includes physical therapy, nonsteroidal anti-inflammatory medicine, cortizone injections, or hyaluronic acid injections.

    1. Treatment failure is indicated by Subjects having symptoms of knee pain, swelling, and trouble with activities for at least 4 to 6 weeks. Subjects would only be enrolled if they fail conservative treatment. Usually physical therapy is administered initially for 6 weeks along with an NSAID medication. If that fails, which means that pain and swelling and disability continue, then injection therapy with corticosteroid or hyaluronic acid (HA) is given. Usually the injection is followed up in 6 to 8 weeks post-injection. If that fails, then Orthobiologics will be discussed (at about 4 to 6 months after treatment).
    2. The subject must fail at least two conservative treatments, which could include physical therapy and NSAIDs, or physical therapy and injections, or NSAIDs and injections.
11. Subjects must have WOMAC and VAS scores of ≥30 and ≥4, respectively at least 2 weeks prior to enrollment.
12. Male and female subjects of reproductive potential must agree to refrain from sexual activity or use effective birth control for a duration of one week before and three months after initiation of treatment with either active treatment modality.
13. Subjects with basal cell, in situ carcinoma, or remote history (i.e., > 3 years ago) history of low-grade cancers (e.g., breast) that were effectively treated may be included.

Exclusion Criteria:

1. Tibia on femur subluxation greater than 1mm. Varus or valgus number greater than 9°.
2. Intra-articular injection to affected knee within 6 weeks of BMA injection
3. Subjects who have had recent administration of intra- articular injection (e.g. corticosteroid, viscosupplement, platelet-rich plasma (PRP), or any other stem cell therapy) within the last 3 months prior to the experimental therapy.
4. Subjects who have had recent systemic (oral (PO), intravenous (IV) and/or intramuscular (IM) within 6 weeks of treatment) administration of corticosteroids; including subjects who are likely to need or who are currently on systemic steroids (e.g., asthma)
5. Subjects with a BMI of >40 and <18 will be excluded.
6. Fever, active infection and ongoing infectious diseases, including HIV and hepatitis
7. Clinically significant diabetes (HGB A1C >7%), cardiovascular (stable cardiovascular (CV) disease as indicated by treating cardiologist within 30 days of enrollment and/or an ejection fraction of <55%), hepatic (Pugh score of Class A or less than 6), or renal disease (Stage 1 or more severe).
8. Malignancy of the blood such as leukemia or lymphoma or those malignancies which are not > 5 years post treatment including prostate cancer, breast cancer, thyroid cancer, kidney cancer or lung cancer. Subjects with an active malignancy, or subjects with a history of any malignancy (e.g., including in situ, basal cell, etc.) will be excluded.
9. Use of anti-rheumatic medications, including methotrexate and other anti-metabolites.
10. Patients that are chronically taking Plavix, Coumadin and other anticoagulants for stroke/myocardial infarction/thromboembolic phenomena prevention, and/or Pradaxa, Xarelto, Mylanta, Fish Oil, Elmiron, Cipro, Levaquin, Quinolones, Ibuprofen, aspirin, Naproxen, CBD oil, Turmeric, or Meloxicam.
11. Current chemo or radiation therapy
12. Current drug or alcohol use disorder
13. Subjects with h/o noncompliance or serious emotional disabilities, and/or any thought disorder, etc. will be excluded
14. History of severe anemia or bleeding disorders (infectious arthritis, hemophilic arthropathy, Charcot's knee) (Anemia for the study is defined as Hgb 12 g/dL.)
15. History of severe metabolic bone disease (osteoporosis, osteomalacia, rickets, osteitis fibrosa cystica, Paget's disease of bone) (Metabolic bone disease is osteoporosis diagnosed by DEXA scan, Leukemia, aplastic anemia or bone Metastasis.)
16. Pregnant or currently breast-feeding. Males and females of reproductive potential will refrain from sexual activity or use effective birth control for up to 90 days following product administration.
17. History of systemic chondrocalcinosis.
18. Vitamin D levels < 30 ng/mL.
19. Subjects who are unwilling to forgo pain medication during and for a 2 weeks before clinical assessments will be excluded to decrease the potential for confounding of the efficacy assessments.
20. Subjects with claudication and vascular disorders (such as varicose veins or peripheral arterial disease), neurological disorders or other disabilities aside from osteoarthritis that may affect ambulation.
21. Physical Exam findings include severe peripheral vascular disease, deep vain thrombosis (DVT), heart murmur, clubbing, open wounds, and other specific knee findings including significant varus or valgus deformity or subluxation of the femoral - tibial joint space, patellar tracking issues, trendelenburg gait or extremity weakness or significant peripheral neuropathy.
22. Subjects may not have popliteal Baker's cyst(s).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Western Ontario McMaster University Osteoarthritis Index (WOMAC) at 3 months | 3 months
  The Western Ontario and McMaster Universities Osteoarthritis Index is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The minimum clinically important difference (MCID) for this parameter is ≥ 10.
Change from Baseline Western Ontario McMaster University Osteoarthritis Index (WOMAC) at 6 months | 6 months
  The Western Ontario and McMaster Universities Osteoarthritis Index is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The minimum clinically important difference (MCID) for this parameter is ≥ 10.
Change from Baseline Western Ontario McMaster University Osteoarthritis Index (WOMAC) at 12 months | 12 months
  The Western Ontario and McMaster Universities Osteoarthritis Index is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The minimum clinically important difference (MCID) for this parameter is ≥ 10.
Change from Baseline Visual Analog Score (VAS) at 3 months | 3 months
  The pain VAS is a unidimensional scale of pain that is widely used and well validated in diverse groups of adult patients. The horizontal scale will be anchored by "no pain" (0) with "worst imaginable pain" (10) being at the opposite extreme. The minimum clinically important difference (MCID) for this measure is VAS ≥ 2
Change from Baseline Visual Analog Score (VAS) at 6 months | 6 months
  The pain VAS is a unidimensional scale of pain that is widely used and well validated in diverse groups of adult patients. The horizontal scale will be anchored by "no pain" (0) with "worst imaginable pain" (10) being at the opposite extreme. The minimum clinically important difference (MCID) for this measure is VAS ≥ 2
Change from Baseline Visual Analog Score (VAS) at 12 months | 12 months
  The pain VAS is a unidimensional scale of pain that is widely used and well validated in diverse groups of adult patients. The horizontal scale will be anchored by "no pain" (0) with "worst imaginable pain" (10) being at the opposite extreme. The minimum clinically important difference (MCID) for this measure is VAS ≥ 2
Magnetic Resonance Imaging (MRI) Evaluation | Baseline and 12 months
  Magnetic resonance imaging (MRI) is a medical imaging technique used in radiology to form pictures of the anatomy and the physiological processes of the body in both health and disease. MRI scanners use strong magnetic fields, radio waves, and field gradients to generate images of the inside of the body.

SECONDARY OUTCOMES:
Change from baseline measure of Fall Risk Functional Testing at 3 months | 3 months
  Fall Risk Functional Testing
Change from baseline measure of Fall Risk Functional Testing at 6 months | 6 months
  Fall Risk Functional Testing
Change from baseline measure of Fall Risk Functional Testing at 12 months | 12 months
  Fall Risk Functional Testing
Change from baseline measure of Frailty Functional Testing at 3 months | 3 months
  Frailty Functional Testing
Change from baseline measure of Frailty Functional Testing at 6 months | 6 months
  Frailty Functional Testing
Change from baseline measure of Frailty Functional Testing at 12 months | 12 months
  Frailty Functional Testing
Change from baseline measure of Joint Specific Range of Motion Functional Testing at 3 months. | 3 months
  Joint Specific Range of Motion Functional Testing
Change from baseline measure of Joint Specific Range of Motion Functional Testing at 6 months. | 6 months
  Joint Specific Range of Motion Functional Testing
Change from baseline measure of Joint Specific Range of Motion Functional Testing at 12 months. | 12 months
  Joint Specific Range of Motion Functional Testing
Change from baseline measure of Obesity Functional Testing at 3 months | 3 months
  Obesity Functional Testing
Change from baseline measure of Obesity Functional Testing at 6 months | 6 months
  Obesity Functional Testing
Change from baseline measure of Obesity Functional Testing at 12 months | 12 months
  Obesity Functional Testing

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Scarpone, D.O., Principal Investigator — Next Generation Regenerative Medicine LLC; James G Unnerstall, Study Director — Next Generation Regenerative Medicine LLC
Locations (3):
- United States (3):
  - Bluetail Medical Group, Chesterfield, Missouri
  - Scarpone Sports Regenerative, Steubenville, Ohio
  - Albano Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
IPD Sharing Plan: Not Applicable